CLINICAL TRIAL: NCT00071838
Title: Zenapax (Daclizumab) Admin to Pts With Multiple Sclerosis (ZAP MS): Effect of Intravenously Admin Humanized Monoclonal Antibody Against the Interleukin-2 Receptor Alpha Subunit (Daclizumab) on Inflammatory Activity in the Central Nervous System
Brief Title: Zenapax (Daclizumab) to Treat Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Bibiana Bielekova, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040019; 04-N-0019
Record Dates: First submitted 2003-10-31; First posted 2003-11-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-16

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Neuroimmunology; Therapy; Demyelinating Disease; Immunological Mechanism; MRI; Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Demyelinating Diseases; Multiple Sclerosis | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will examine the safety of Zenapax (daclizumab) in patients with multiple sclerosis (MS). MS is thought to be caused by an over-reactive immune response. T-lymphocytes (cells of the immune system), are thought to damage myelin, a substance that covers the nerve and parts of the spinal cord and is damaged in patients with MS. Interleukin-2 is a natural substance in the body that is necessary for the growth of T-lymphocytes. Zenapax is a genetically engineered antibody that blocks the activity of interleukin-2 and thus interferes with the growth of lymphocytes. Therefore, Zenapax may prevent some of the damage to myelin that occurs in multiple sclerosis.

Patients between 18 and 65 years of age with relapsing remitting MS may be eligible for this study. Patients with secondary-progressive or primary progressive MS may not participate. Candidates will be screened with a complete neurological and medical evaluation and review of medical records.

Participants will undergo the following tests and procedures:

* Baseline evaluation: Participants have four magnetic resonance imaging (MRI) scans over a 3-month period to assess disease activity. For the MRI scans, the patient lies on a table that slides into the scanner - a narrow metal cylinder with a strong magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Only patients with activity at or above a certain level are eligible to continue with the treatment phase of the study.
* Zenapax treatment: Patients receive intravenous (through a vein) infusions of Zenapax. The first two infusions are 2 weeks apart, followed by 13 monthly infusions.
* MRI scans: Patients undergo MRI scanning before every infusion to evaluate disease activity and identify new brain lesions.
* Blood and urine tests: Blood and urine samples are collected at each clinic visit for routine laboratory evaluations, immunologic study, and genetic testing to determine a predisposition for responding to Zenapax treatment.
* Lumbar puncture (spinal tap): This procedure will be done during the last month before starting treatment and during the seventh month of treatment to examine immune changes that occur in the cerebrospinal fluid (CSF), which circulates through and surrounds the brain and spinal cord. A local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Skin test: A needle is placed just under the skin is done to assess the patient's immune status to common antigens such as tetanus, mumps and candida.
* Lymphocytopheresis: Lymphocytes are collected three times - once during the last month of baseline before starting treatment, once during the fifth month of treatment, and once during the last month of treatment - for immunologic study. Blood is collected through a needle in an arm vein in a similar way to donating blood. The blood flows from the vein through a catheter (plastic tube) into a machine that separates it into its components by centrifugation (spinning). The lymphocytes are removed and the rest of the blood (red cells, plasma and platelets) is returned to the body, either through the same needle or through another needle in the other arm.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is considered a T cell-mediated autoimmune disease leading to central nervous system (CNS) inflammation, demyelination, axonal loss, and leads to substantial disability in young adults. Existing approved treatments include interferon beta, glatiramer acetate and mitoxantrone. These therapies are only moderately effective in reducing disease activity.

The Neuroimmunology Branch (NIB) has during the last three years tested the tolerability and safety of monthly intravenously administered daclizumab (Zenapax(Registered Trademark)), a humanized monoclonal antibody against the IL-2 receptor alpha chain, in patients who receive interferon-beta, but responded incompletely to therapy with interferon-beta. Daclizumab has been well tolerated and inhibited inflammatory disease activity by almost 90%. Under an amendment of this protocol, it was demonstrated that the efficacy of daclizumab is maintained once interferon-beta therapy is discontinued.

In the current trial, we will test the efficacy of daclizumab alone in relapsing-remitting MS patients. This trial is a single-centre, open-label, baseline to treatment cross-over phase II trial. Daclizumab will be administered intravenously at 1mg/kg bodyweight. Contrast-enhancing MRI lesions will serve as the primary outcome measure in this phase II trial, and a number of clinical, MRI, and immunological parameters will be measured as secondary and tertiary outcomes. Daclizumab is a promising new immunomodulatory treatment for relapsing-remitting MS.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PRE-TREATMENT SCREENING:

To be eligible for entry into the study, patients must meet the following criteria at the time of enrollment. Re-assessment of the inclusion criteria will occur on day zero of the twelve-month treatment phase.

Between the ages of 18 and 65 years, inclusive.

Patients with relapsing-remitting MS according to published criteria.

EDSS score between 1.0 and 5.5.

Patients have either failed standard therapies (interferon-beta, glatiramer acetate) by clinical measures, or are not eligible for standard therapies, or opted not to start or continue with any of the standard therapies.

Patients are able to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care.

Age criteria for inclusion in this study follow those of published diagnostic criteria for multiple sclerosis. Due to the uncommon occurrence of MS in individuals under the age of 18 and the requirement to study a large MS cohort to include these rarely occurring patients, this is an appropriate lower age range.

Patient decision not to start, or not to continue with standard immunomodulatory therapy, has to be made by the patient after discussing conventional treatment options to ensure the patient has made an informed decision. Additionally, the consent document provided to the patient will explicitly state the currently approved therapies and their potential benefits.

ELIGIBILITY CRITERIA FOR INITIATING THERAPY:

To be eligible to proceed to the treatment phase of the study, patients must have at least two new gadolinium-enhancing lesions or greater in the four sequential baseline MRI scans (average of greater than or equal to 0.5 gadolinium-enhancing lesions or more).

Patients can not have a relapse during 30 days before initiation of treatment. If a relapse occurs during this period and eligibility criteria are otherwise fulfilled, treatment (day one) will be delayed while corticosteroids are administered. If corticosteroids are administered, the MRI during that period will not be considered. An additional MRI will be added at 4 weeks following the completion of corticosteroids, to maintain a total of four MRI's that are analyzed in the baseline period. In the event of relapse, the baseline period will be prolonged, as necessary, to meet these criteria.

EXCLUSION CRITERIA FOR PRE-TREATMENT SCREENING:

Patients will be excluded from the study if any of the exclusion criteria exist at the time of enrollment. Re-assessment of the exclusion criteria will occur on day zero of the twelve month treatment phase.

MEDICAL HISTORY:

Diagnosis of secondary-progressive or primary-progressive MS, as defined by published diagnostic criteria.

Abnormal screening/baseline blood tests exceeding any of the limits defined below:

* Serum alanine transaminase or aspartate transaminase levels which are greater than three times the upper limit of normal values.
* Total white blood cell count less than 3000/mm(3)
* Platelet count less than 85000/mm(3)
* Serum creatinine level greater than 2.0 mg/dl
* Serological evidence of HIV or active hepatitis A, B or C infection since the effects of daclizumab are not defined in these patients
* Positive pregnancy test

Pregnant or breast-feeding female.

History or signs of immunodeficiency.

Concurrent clinically significant (as determined by the investigators) cardiac, immunological, pulmonary, neurological, renal or other major disease.

Any contraindication to monoclonal antibody therapy. Contraindication to monoclonal antibody therapy includes prior history of serum-sickness or similar hypersensitivity reaction to receipt of monoclonal antibody or intravenous immunoglobulin therapies.

Patients with cognitive impairments who are unable to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care.

TREATMENT HISTORY:

If prior treatments were administered, the patient must be off the following treatment agents for the required period prior to enrollment:

* Glatiramer acetate, interferon-beta - 24 weeks
* IVIg, azathioprine, methotrexate, cyclophosphamide, mitoxantrone, plasma exchange, cyclosporine, oral myelin, cladribine and other immunosuppressive treatments - 24 weeks
* Corticosteroids - 6 weeks

Prior treatment with other investigational drugs or procedures will be evaluated individually by the investigators.

MISCELLANEOUS EXCLUSIONS:

History of alcohol or drug abuse within the 5 years prior to enrollment.

Female patients who are not post-menopausal or surgically sterile who are not using an acceptable method of contraception. Acceptability of various methods of contraception will be at the discretion of the investigator. Documentation that the patient is post-menopausal or surgically sterile must be available prior to enrollment.

Male patients who are not surgically sterile and not practicing adequate contraception. Acceptability of various methods of contraception will be at the discretion of the investigator. Documentation that the patient is surgically sterile must be available prior to enrollment.

Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the patient returning for follow-up visits on schedule.

Previous participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-10-30; Primary Completion 2007-10-04 (Actual); Study Completion 2011-08-16 (Actual)

PRIMARY OUTCOMES:
Reduction in mean number of new gaolinium-enhancing lesions in the treatment phase (Weeks 18 to 30) versus baseline (Weeks -12 to 0).

SECONDARY OUTCOMES:
Mean change in the MS functional composite from completion of treatment. Reduction of mean number of new gaolinium-enhancing lesions at the completion of treatment. Mean change in Multiple Sclerosis Quality of Life Inventory from completion of t...

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Martin R, McFarland HF, McFarlin DE. Immunological aspects of demyelinating diseases. Annu Rev Immunol. 1992;10:153-87. doi: 10.1146/annurev.iy.10.040192.001101. PMID 1375472
- [Background] Wucherpfennig KW, Strominger JL. Molecular mimicry in T cell-mediated autoimmunity: viral peptides activate human T cell clones specific for myelin basic protein. Cell. 1995 Mar 10;80(5):695-705. doi: 10.1016/0092-8674(95)90348-8. PMID 7534214
- [Background] Gran B, Hemmer B, Vergelli M, McFarland HF, Martin R. Molecular mimicry and multiple sclerosis: degenerate T-cell recognition and the induction of autoimmunity. Ann Neurol. 1999 May;45(5):559-67. doi: 10.1002/1531-8249(199905)45:53.0.co;2-q. PMID 10319877